CLINICAL TRIAL: NCT05073562
Title: A Study on the Effectiveness of IFA Supplementation, Deworming, and Nutrition Education in Addressing Anemia Among Adolescent Girls in Two Counties in Liberia
Brief Title: Nutrition Intervention to Address Anemia Among Adolescent Girls in Liberia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in funding availability
Sponsor: Boston Children's Hospital (Other)
Collaborators: UNICEF (Other); Ministry of Health, Liberia (Other); Liberia Institute of Statistics and Geo-Information Services (Unknown)
Responsible Party: Principal Investigator, Julia Rubin-Smith, Global Health Faculty/Assistant in Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P00036604
Record Dates: First submitted 2021-08-01; First posted 2021-10-11 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Nutritional Anemia; Nutritional Deficiency; Iron Deficiency Anemia Treatment; Folic Acid Deficiency Anemia, Dietary; Adolescent Development; Knowledge, Attitudes, Practice; Food Habits
MeSH Terms: conditions — Malnutrition; Behavior; Feeding Behavior | interventions — Iron; Folic Acid; Dietary Supplements; Mebendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrition+ Intervention (Experimental): This group will receive a structured nutrition education package provided by Community Health Assistants (CHAs) based on a handbook on nutrition education developed by UNICEF with collaboration from the Liberia Ministry of Health. The structured nutrition education package will focus on four key areas: causes and prevention of anemia, healthy eating and food choices, hand washing, and physical exercise. Participants in the intervention group will also receive IFA supplementation on a weekly basis for the duration of the study, and a one-time oral deworming treatment (mebendazole), which will be administered once at the beginning of the study.
  Interventions: Dietary Supplement: Iron and folic acid (IFA) supplementation; Behavioral: Targeted nutrition education; Drug: Mebendazole Pill
- Control group - standard services only (Active Comparator): This group will receive only the current package of basic nutrition services provided at the health facility and at community level by health workers and CHAs, respectively.
  Interventions: Other: Standard nutrition services

INTERVENTIONS:
Dietary Supplement: Iron and folic acid (IFA) supplementation — Weekly IFA supplementation for duration of the study.
  Arms: Nutrition+ Intervention
Behavioral: Targeted nutrition education — Structured nutrition education package delivered at household level by trained Community Health Assistants (CHAs)
  Arms: Nutrition+ Intervention
Drug: Mebendazole Pill — One-time deworming treatment with mebendazole.
  Arms: Nutrition+ Intervention
Other: Standard nutrition services — Basic nutrition services currently provided at the health facility and at community level in Liberia
  Arms: Control group - standard services only

SUMMARY:
The purpose of this study is to evaluate the feasibility and effectiveness of weekly iron and folic acid (IFA) supplementation and one-time deworming treatment at the community level in improving hemoglobin levels among adolescent girls in Liberia, West Africa, and to assess the feasibility and effectiveness of a targeted nutrition education program in improving nutrition knowledge, attitudes, and practices in the same population.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girl aged 10 - 19 years at the time of enrollment
* Lives within the selected study communities in Montserrado or Margibi counties
* Caregiver/adolescent consents to participate in the study

Exclusion Criteria:

* Currently pregnant
* Active malaria infection as defined by positive rapid diagnostic test (RDT)
* Severe acute malnutrition at the time of enrollment
* Known malignancy
* Known sickle cell disease

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Will enroll females, assessed by participant self-identification
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in participants' hemoglobin level from enrollment to completion of the study | Baseline and Week 12
  Point of care hemoglobin testing will be conducted at enrollment and at the conclusion of the study.

SECONDARY OUTCOMES:
Changes in responses to questions in the Nutrition Knowledge, Attitudes, and Practice (KAP) survey from baseline to follow up evaluation | Baseline and Week 12
  Increase in nutrition-related knowledge, and improvements in nutrition practices as evidenced by changes in responses to the KAP survey, which is based on validated measures of nutrition-related knowledge, attitudes, and practices, and has been modified for appropriateness to the target population of this study.
Feasibility of targeted intervention for scale-up to country-wide enhanced nutrition services | 12 weeks
  Successful completion of study visits by Community Health Assistants, specifically ability to conduct every scheduled visit without skipping visits or households, within the timeframe of scheduled work day.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rubin-Smith, MD, MSPH, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No